CLINICAL TRIAL: NCT00832026
Title: Trans Nasal Insufflation for the Treatment of Snoring and Obstructive Sleep Apnea
Brief Title: Trans Nasal Insufflation for the Treatment of Snoring
Acronym: TNI
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00019483
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2018-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; snoring; sleep apnea treatment; TNI; Trans nasal insufflation; Open CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep apnea: Patients with diagnosed obstructive sleep apnea
  Interventions: Device: Trans Nasal Insufflation (TNI) [nasal canula]

INTERVENTIONS:
Device: Trans Nasal Insufflation (TNI) [nasal canula] — Trans Nasal Insufflation, or TNI, uses air at flow rates delivered through a small nasal canula to reduce the severity and frequency of sleep apnea events.
  By using TNI we hope to increase the amount of air that the patient can breathe during periods of obstructive sleep disordered breathing.

SUMMARY:
This research is being done to examine if a nasal cannula can be used to keep the throat open during sleep, thereby treating sleep apnea.

People with sleep apnea and people who snore without sleep apnea may take part in this study. Sleep apnea is a disorder caused by pauses in breathing due to repetitive closure of the throat. The most common form of treatment for sleep apnea is continuous positive airway pressure (CPAP) therapy. While CPAP therapy remains the simplest and most effective treatment for snoring and sleep apnea, patients have to wear a nasal mask throughout the night. For this reason, patients often have difficulty sticking to therapy.

Participants enrolled in this study will spend 3-nights in a sleep laboratory. In all nights, the investigators will monitor your sleep and your breathing throughout the night. The investigators will apply several electrodes (sensors) to your scalp and face to monitor your sleep and breathing, and other sensors to your chest, abdomen, cheek, and a finger to monitor your breathing and oxygen level.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults over the age of 21
* Diagnosed obstructive sleep apnea

Exclusion Criteria:

* Unstable cardiovascular disease
* Uncontrolled hypertension (BP > 190/110)
* Severe intrinsic lung diseases (supplemental O2 > 2 L/min during the day)
* History of chronic renal insufficiency
* History of hepatic insufficiency
* Pregnancy
* Bleeding disorders or Coumadin use
* Sleep Disorders other than Obstructive Sleep Apnea (OSA)
* Tracheostomy
* Allergy to lidocaine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with obstructive sleep apnea are eligbile to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2004-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in inspiratory airflow | 2 nights

SECONDARY OUTCOMES:
Change in sleep apnea severity (AHI) | 2 nights
Change in Ratio of apnea-to-hypopnea events | 2-nights

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Result] McGinley BM, Patil SP, Kirkness JP, Smith PL, Schwartz AR, Schneider H. A nasal cannula can be used to treat obstructive sleep apnea. Am J Respir Crit Care Med. 2007 Jul 15;176(2):194-200. doi: 10.1164/rccm.200609-1336OC. Epub 2007 Mar 15. PMID 17363769